CLINICAL TRIAL: NCT03246672
Title: Development of a Weight Maintenance Intervention for Bariatric Surgery Patients
Acronym: MAINTAIN-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPO 16-331
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-07

CONDITIONS: Obesity, Morbid
Keywords: obesity, morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: All participants receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- maintenance (Experimental): behavioral intervention to increase adherence to lifestyle recommendations
  Interventions: Behavioral: maintenance intervention

INTERVENTIONS:
Behavioral: maintenance intervention — Participants will receive calls at weeks 1, 2, 3, 4, 6, 8, 10, 12, and 14 that focus on satisfaction with outcomes of behavior change, self-monitoring, relapse planning, and social support.

SUMMARY:
Although bariatric surgery is highly effective for inducing significant weight loss and resolution of comorbidities, weight regain following surgery is a common problem. This pilot study will test the feasibility and acceptability of an intervention designed to help bariatric surgery patients maintain weight loss. Findings from this pilot will provide the foundation for a randomized controlled trial to evaluate the efficacy of the intervention.

DETAILED DESCRIPTION:
The first intervention telephone call will occur one week following the baseline assessment. Calls will be made weekly in the first month (weeks 1, 2, 3, 4) and biweekly calls during months 2-4 (weeks 6, 8, 10, 12, 14). The goal of this intervention is to increase adherence to recommendations that patients are already receiving from their bariatric team as part of standard of care. Thus, each call will address maintenance skill building and anticipatory problem solving based on the processes outlined in the investigators' conceptual model and operationalized in the investigators' previous weight loss maintenance protocol. Relapse prevention planning will help patients identify situations in which overeating is common in the bariatric population (e.g., loss of control eating related to emotions, disinhibition).

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery at a participating VA site
* Laparoscopic Roux-en-Y gastric bypass (RYGB) or laparoscopic vertical sleeve gastrectomy (SG) six to 18 months prior to the time of data pull
* English as preferred language
* Regular access to a telephone

Exclusion Criteria:

* Receipt of procedure to prevent gastric cancer
* Revisional bariatric surgery
* Hearing impairment
* Cancer not in remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine I. Voils, PhD, Principal Investigator — William S. Middleton Memorial Veterans Hospital, Madison, WI
Locations (1):
- William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adamek KE, Ramadurai D, Gunzburger E, Plomondon ME, Ho PM, Raghavan S. Association of Diabetes Mellitus Status and Glycemic Control With Secondary Prevention Medication Adherence After Acute Myocardial Infarction. J Am Heart Assoc. 2019 Feb 5;8(3):e011448. doi: 10.1161/JAHA.118.011448. PMID 30712488
- [Derived] Voils CI, Adler R, Strawbridge E, Grubber J, Allen KD, Olsen MK, McVay MA, Raghavan S, Raffa SD, Funk LM. Early-phase study of a telephone-based intervention to reduce weight regain among bariatric surgery patients. Health Psychol. 2020 May;39(5):391-402. doi: 10.1037/hea0000835. Epub 2020 Jan 30. PMID 31999175

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from January to March 2018. These participants were identified using electronic medical record data indicating that they had bariatric surgery for weight loss at one of four VA hospitals: West Roxbury, MA; Long Beach, CA; Palo Alto, CA; and Ann Arbor, MI.
Pre-assignment Details: 33 participants provided verbal consent. Of those, 3 were unable to be reached and 30 were reached by telephone to complete baseline measures and were scheduled for their first intervention phone call. Of those 30, 29 participants were reached for the first intervention phone call, and 1 participant unable to be reached for further participation.
Period: Overall Study
Arm/Group | Maintenance
Started | 30
Completed First Phone Call | 29
Completed | 28
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 30 participants completed baseline measures.
Arm/Group | Maintenance
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 22
  More than one race | 2
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Percentage of contacted patients who consent to be in the study
Time Frame: week 0
Population: # of patients for whom phone screening was attempted
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance
Number analyzed (Participants) | 69
Participants | 33

2. Primary Outcome: Retention Rate
Description: Percentage of patients with baseline data who complete 16-week outcome assessments
Time Frame: 16-week outcome assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance
Number analyzed (Participants) | 30
Participants | 28

3. Secondary Outcome: Weight
Description: Patient weight obtained from the electronic medical record on the clinical visit date closest to the 16-week study assessment date
Time Frame: 16 weeks
Population: The N=30 is based on the number of participants who provided baseline data according to Intent-to-treat principles
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Maintenance
Number analyzed (Participants) | 30
pounds | 213.7 (43.1)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Adverse events were volunteered by participants during intervention or assessment phone calls; they were not systematically queried in this minimal-risk intervention.
Arm/Group | Maintenance
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT03246672/Prot_SAP_000.pdf